CLINICAL TRIAL: NCT03969771
Title: A Mindfulness Based Intervention as a Key Component of Successful Workplace Functioning and Personal Well-being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Workers Compensation Board of Manitoba (Unknown); Catholic Health Corporation of Manitoba (Unknown)
Responsible Party: Principal Investigator, Michael McIntyre, Principal Investigator, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2018:467
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Emotional Stress; Work Related Illnesses; Burnout, Professional; Burnout Syndrome
Keywords: Mindfulness-Based Stress Reduction; Mindfulness
MeSH Terms: conditions — Stress, Psychological; Burnout, Professional; Burnout, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: 2 x 2 Mixed Factorial Design, with Group (frequently absent / control) as the between-subjects factor and Time (pre / post) as the within-subjects factor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frequently Absent (Experimental): 8 weeks of training in Mindfulness-Based Stress Reduction
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Normal Attendees (Controls) (Active Comparator): 8 weeks of training in Mindfulness-Based Stress Reduction
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The MBSR program was developed by the University of Massachusetts Medical School.

SUMMARY:
This study will evaluate the effectiveness of an 8-week program in Mindfulness-Based Stress Reduction (MBSR) in reducing work absences and improving the well-being of healthcare workers. Half of participants will be healthcare employees who are frequently absent from work, whereas the other half will be healthcare employees with normal attendance patterns. All participants will undergo MBSR training and the outcomes of both groups will be evaluated.

DETAILED DESCRIPTION:
The scientific literature is replete with evidence that the demands and pace of providing healthcare is associated with high levels of stress, anxiety, burnout, diminished work engagement, and frequent absence. For example, Actionmarguerite is one of the largest personal care facilities in Western Canada. They have over 500 employees who routinely deal with the task of providing care to a large population of individuals requiring high levels of support. A great many of the residents are suffering progressive dementia and some have very difficult behavioural issues. Caretaker stress is exacerbated by the fact that even the highest, most compassionate levels of care are not likely to result in improvement. The employee population is, therefore, taxed such that one might expect to observe a high level of stress-related illness and accidents. An internal examination of the employee database has identified an interesting circumstance. Approximately fifty of the employees have patterns of persistent, recurring injury, show signs of stress/caretaker stress, depletion, and preoccupation. This group has also largely exhausted their sick leave benefits. Clearly, the medical treatments and the time away from work have not cured the underlying predisposition for accidental injury and illness for these individuals. Such may be the case for employees of other healthcare facilities in Canada and elsewhere.

The question has arisen whether Mindfulness Based Stress Reduction (MBSR) as an option available for frequently absent employees would alter the pattern of recurrence and reduce stress. MBSR is a program initially developed at the University of Massachusetts Medical Centre as a means of reducing the chronic stress of patients experiencing high levels of disabling, chronic physical pain. Scientific evaluation of the program demonstrated significant success. Importantly, MBSR training has been shown to reduce stress and anxiety and promote psychological well-being, both for individuals in the general population and for healthcare workers in particular. Indeed, our own work has demonstrated that MBSR resulted in a very substantial and statistically significant reduction of stress in a diverse group of individuals employed in healthcare.

The purpose of the present research is to examine the efficacy of a program of MBSR to interrupt the existing pattern of recurrent work-related accidents, injuries, and illness; and also, to promote both psychological and physical well-being and to allow a more meaningful and successful return to work. We intend to recruit four groups of thirty participants from two local healthcare institutions (Actionmarguerite and St. Amant). Each group will consist of (a) fifteen individuals identified by the respective institutions as frequently-absent employees, and (b) fifteen individuals who express interest in participation and are randomly selected from the general population of healthcare employees at the two institutions to serve as statistical controls. All participants will receive an intervention of MBSR training. They will complete a survey battery both pre- and post- intervention and provide access to their work histories. We hope to establish that MBSR can be an extremely useful component of a program intended to reverse patterns of frequent absence.

ELIGIBILITY:
Inclusion Criteria:

* An employee of Actionmarguerite or St. Amant Centre in Winnipeg, Manitoba, Canada who has contact with patients.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Number of Work Absences | Baseline and 2 years
  A comparison between the number of work absences in the 2 years prior versus 2 years following the intervention. The desired outcome is a statistically significant decrease in the number of work absences.

SECONDARY OUTCOMES:
Change in the Number of Workplace Accidents and Injuries | Baseline and 2 years
  A comparison between the number of workplace accidents and injuries in the 2 years prior versus 2 years following the intervention. The desired outcome is a statistically significant decrease in the number of workplace accidents and injuries.
Change in the Number of Late Work Arrivals | Baseline and 2 years
  A comparison between the number of late work arrivals in the 2 years prior versus 2 years following the intervention. The desired outcome is a statistically significant decrease in the number of late work arrivals.
Change in Perceived Stress | Baseline and 8 weeks
  Assessed by total scores on the Perceived Stress Scale (Cohen et al., 1983), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant decrease in perceived stress.
Change in Burnout | Baseline and 8 weeks
  Assessed by total scores and subscale scores (personal burnout, work burnout, client burnout) on the Copenhagen Burnout Inventory (Kristensen et al., 2005), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant decrease in burnout.
Change in Positive and Negative Emotions | Baseline and 8 weeks
  Assessed by subscale scores (positive affect, negative affect) on the Positive and Negative Affect Schedule (Watson et al., 1988), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in positive emotions and a statistically significant decrease in negative emotions.
Change in Anxiety | Baseline and 8 weeks
  Assessed by total scores on the State-Trait Anxiety Inventory (Spielberger, 1983), which range from 1 to 4 when item scores are averaged. The desired outcome is a statistically significant decrease in anxiety.
Change in Health Locus of Control | Baseline and 8 weeks
  Assessed by subscale scores (internal, chance, powerful others) on the Multidimensional Health Locus of Control Scale (Wallston et al., 1978), which range from 1 to 6 when item scores are averaged. The desired outcome is a statistically significant increase in internal health locus of control.
Change in Workplace Deviance | Baseline and 8 weeks
  Assessed by total scores on the Workplace Deviance Scale (Bennett & Robinson, 2000), which range from 1 to 7 when item scores are averaged. The desired outcome is a statistically significant decrease in workplace deviance.
Change in Mindfulness | Baseline and 8 weeks
  Assessed by total scores and subscale scores on the Five Facet Mindfulness Questionnaire (Baer et al., 2006), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in mindfulness.
Change in Self-Compassion | Baseline and 8 weeks
  Assessed by total scores and subscale scores on the Self-Compassion Scale (Neff, 2003), which range from 1 to 5 when item scores are averaged. The desired outcome is a statistically significant increase in self-compassion.
Change in Fears of Compassion | Baseline and 8 weeks
  Assessed by total scores and subscale scores on the Fears of Compassion Scales (Gilbert et al., 2011), which range from 0 to 4 when item scores are averaged. The desired outcome is a statistically significant decrease in fears of compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McIntyre, Ph.D., Principal Investigator — St. Boniface Hospital Research Centre
Locations (1):
- St. Boniface Hospital Research Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No